CLINICAL TRIAL: NCT00070551
Title: A Phase I Study of GTI2040 (NSC 722929; IND 67368) in Combination With High-dose Cytarabine in Refractory or Relapsed Acute Myeloid Leukemia (AML)
Brief Title: GTI-2040 and High-Dose Cytarabine in Treating Patients With Refractory or Relapsed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01443; 0304; CDR0000334898; OSU-20030030; NCI-6108; OSU-0304; U01CA076576 (NIH)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — GTI2040; Cytarabine

ARMS (2):
- Stratum I (GTI-2040, cytarabine) (Experimental): Patients receive GTI-2040 IV continuously on days 1-6 and high-dose cytarabine IV over 2 hours twice daily on days 2, 4, and 6.
  Interventions: Biological: GTI-2040; Drug: cytarabine; Other: pharmacological study; Other: laboratory biomarker analysis
- Stratum II (GTI-2040, cytarabine) (Experimental): Patients receive GTI-2040 IV continuously on days 1-6 and high-dose cytarabine IV over 4 hours once daily on days 2-6. In both strata, treatment continues in the absence of unacceptable toxicity.
  Interventions: Biological: GTI-2040; Drug: cytarabine; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: GTI-2040 — Given IV
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Other: pharmacological study — Optional correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of GTI-2040 and high-dose cytarabine in treating patients with refractory or relapsed acute myeloid leukemia. GTI-2040 may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth. Drugs used in chemotherapy, such as cytarabine, use different ways to stop cancer cells from dividing so they stop growing or die. Giving GTI-2040 together with cytarabine may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose and recommended phase II dose of GTI-2040 and high-dose cytarabine in patients with relapsed or refractory acute myeloid leukemia.

SECONDARY OBJECTIVES:

I. Determine the therapeutic response in patients treated with this regimen. II. Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a dose-escalation study. Patients are stratified according to age (under age 60 vs age 60 and over). Patients are assigned to 1 of 2 strata.

Stratum I (under age 60): Patients receive GTI-2040 IV continuously on days 1-6 and high-dose cytarabine IV over 2 hours twice daily on days 2, 4, and 6.

Stratum II (age 60 and over): Patients receive GTI-2040 IV continuously on days 1-6 and high-dose cytarabine IV over 4 hours once daily on days 2-6.

In both strata, treatment continues in the absence of unacceptable toxicity.

Cohorts of 3-6 patients per stratum receive escalating doses of GTI-2040 and high-dose cytarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 6-51patients will be accrued for this study within 2-16 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed acute myeloid leukemia according to the WHO classification
* Relapsed or refractory disease, meeting 1 of the following criteria:

  * Unresponsive to initial treatment
  * Recurrent disease after treatment with prior conventional or high-dose chemotherapy with or without stem cell support
* CNS involvement allowed provided there are no residual leukemic cells detected in the cerebrospinal fluid after intrathecal or radiation chemotherapy
* Performance status - ECOG 0-2
* At least 4 weeks
* Bilirubin no greater than 2 times upper limit of normal* (ULN) (unless due to Gilbert's syndrome)
* AST and ALT no greater than 3 times ULN*
* Creatinine no greater than 1.5 mg/dL*
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Resting ejection fraction at least 50%*
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergy to study medications
* No ongoing or active infection requiring IV antibiotics
* No other concurrent uncontrolled illness
* No serious medical or psychiatric illness that would preclude giving informed consent
* More than 4 weeks since prior chemotherapy (except hydroxyurea) (6 weeks for nitrosoureas or mitomycin)
* No other concurrent chemotherapy
* No concurrent hormonal therapy except steroids for adrenal failure and hormones for non-disease-related conditions (e.g., insulin for diabetes)
* More than 4 weeks since prior radiotherapy
* No concurrent palliative radiotherapy
* Prior therapy with antisense oligonucleotides allowed provided no toxic effects were experienced that were directly attributable to the antisense agents
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent chronic systemic anticoagulant therapy for medical conditions (e.g., prior deep vein thrombosis or atrial fibrillation)

  * Concurrent heparin to maintain central line patency (i.e., catheter flush) is allowed
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2003-09; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to day 42

SECONDARY OUTCOMES:
Therapeutic response | Up to 6 years
  Standard paired statistical tests, parametric and nonparametric, will be used to baseline with treatment values. With data collected serially over time, repeated measures analysis of variance will be used to analyze data.
Change in R2 expression in circulating and marrow leukemia cells | From baseline to up to 6 years
  Standard paired statistical tests, parametric and nonparametric, will be used to baseline with treatment values. With data collected serially over time, repeated measures analysis of variance will be used to analyze data.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Marcucci, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States